CLINICAL TRIAL: NCT02945306
Title: Does Sleep Disordered Breathing in Pre School Age Children Cause Cognitive Weakness Reversible by Adenotonsillectomy? A Feasibility Study
Brief Title: Sleep Disordered Breathing, Adenotonsillectomy, Cognition and Pre-school Age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Principal Investigator, Mike Tremlett, Consultant Anaesthetist, South Tees Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016048
Record Dates: First submitted 2016-07-29; First posted 2016-10-26 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Sleep Disordered Breathing
Keywords: Sleep Disordered Breathing; Adenotonsillectomy; Child
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Watchful Waiting; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adenotonsillectomy (Experimental): Removal of tonsils and adenoids under a general anaesthetic
  Interventions: Procedure: Adenotonsillectomy
- Watchful waiting with supportive care (Active Comparator): Reassurance with active medical treatment of conditions associated with Sleep Disordered Breathing such as otitis media with effusion and allergic rhinitis
  Interventions: Drug: Watchful waiting with supportive care

INTERVENTIONS:
Procedure: Adenotonsillectomy
  Arms: Adenotonsillectomy
Drug: Watchful waiting with supportive care — Use of widely prescribed medicines to treat associated conditions
  Arms: Watchful waiting with supportive care

SUMMARY:
Sleep disorder breathing (SDB) is a condition affecting 10% of children aged 2-6 years. It is a combination of snoring most nights during sleep, patchy sleep, short periods of stopping breathing (apnoea) and usually big tonsils. Most of these children get better with no treatment by 8 years old. It has been suggested that having SDB mean that some children concentrate and behave less well during the day and may learn more slowly than children who don't snore. It has become common for many Ear, Nose and Throat (ENT) surgeons to take out tonsils and adenoids (adenotonsillectomy) for this condition. Removing the tonsils and adenoids (which are normally big at this age) means that most children quickly stop snoring and seem to be cured. Unfortunately it is not clear if this operation makes any difference to learning compared to just watching the child and letting them "grow out" of the condition (watchful waiting).

There is no set treatment in the UK today. Children may be offered adenotonsillectomy or watchful waiting; it is not know which, long term, is the right thing to do. Therefore the investigators wish to do a study looking at these two different treatments to see if there is a difference in children's learning over time between the two different treatments. The investigators will look at children with SDB, measure their learning (and behaviour) and then randomly select which children get one treatment or the other. They will then re-measure learning (and behaviour) 7 months later to see if there is any difference between the two groups. The investigators will also scientifically measure their sleep. This is possibly quite a difficult study to do, the investigators are unsure whether families will agree to take part and how easy it will be to measure learning with such young children (aged 2:6 - 5).

DETAILED DESCRIPTION:
Purpose and Design. Large numbers of children snore on a regular basis in UK. It is known that habitual snoring is associated with cognitive weakness but not known if it is the cause of cognitive weakness. Teenagers who snored at a young age do less well at school than peers, who did not snore at a young age, but it is not known if this is due to the snoring or multiple other confounding factors.

More than 60% of children who snore regularly at 3 years of age have stopped regularly snoring by 7 years of age. They grow out of SDB with no active treatment. If their tonsils and adenoids are removed 80% will immediately stop snoring (and will be cured). Research shows that if tonsils and adenoids are removed at 6-8 years old, there is no difference in cognitive abilities between the group who had adenotonsillectomy and those that did not.

It is not known if several years of habitual snoring, sleep fragmentation and recurrent short-lived episodes of hypoxia cause minor changes to the developing brain causing cognitive weakness. Therefore it is not known if taking tonsils and adenoids out at a young age (2-4 years) when they first start snoring, thus avoiding several years of habitual snoring, sleep fragmentation and recurrent mild hypoxia, makes a difference to cognition in the future. It is not known if a period of a number of years of habitual snoring (with possible sleep fragmentation and recurrent episodes of hypoxia) causes irreversible cognitive weakness, reversible cognitive weakness or no cognitive weakness at all.

35,000 children undergo adenotonsillectomy in England and Wales per year with the second most common indication being SDB (habitual snoring and other features of recurrent upper airway obstruction).

The balance of benefits versus detrimental effects of adenotonsillectomy in children with SDB is not accurately known. The detrimental effects are well known. They include significant pain for at least 7 days for most children, bleeding after the operation in 1%, and very, very rarely death. The benefits are less clear. Adenotonsillectomy in pre-school age children with SDB results in improved behaviour and quality of life scores in the short term but it is not known if there is an effect on cognition. The effect of adenotonsillectomy on cognitive development versus the effect of watchful waiting with supportive care (treatment of associated conditions such as chronic otitis media with effusion and rhinitis) needs investigation, if clinicians are to give families a true description of advantages and disadvantages of surgery for SDB.

The investigators therefore need to ask the question - Does adenotonsillectomy in preschool age children alter future cognitive development? Answering this question will require a large, multicentre randomised controlled study.

This study aims to assess the feasibility of carrying out this large randomised control trial. It will try to answer the following questions:

1. Can the investigators effectively measure cognition in preschool age children?
2. Will parents be prepared to take part in such a study?
3. Can the investigators obtain useful sleep studies in these young children at home?
4. Will children stay in the study long enough to allow follow up?
5. Can the investigators define values allowing us to power a larger randomised control trial?
6. Does the SRBD scale work as a pragmatic screening tool for SDB in a UK population? Although numbers in this study will be small, the investigators may find a large difference in outcomes between the two groups making a larger randomised control trial unnecessary. Data from this study will therefore be analysed.

Recruitment:

All children between 2.6 years and 5 years, referred to two ENT surgeons in Middlesbrough by General Practitioners in the Teesside geographical area with possible SDB will be considered for recruitment into the trial. They will be offered entry into the trial if they meet inclusion and exclusion criteria. The aim of these criteria is to have a study population of children with the typical clinical features of SDB that would be actively considered by informed ENT surgeons as possibly being offered adenotonsillectomy as a treatment in typical UK practice.

Clear inclusion and exclusion criteria will be in place to delineate this population.

Randomisation:

Participants will be randomised to one of two treatments, either early removal of tonsils and adenoids under general anaesthesia or watchful waiting, to allow the child to potentially grow out of the condition without surgical intervention.

Consent:

Clear unambiguous information will be provided to the parents/guardians of prospective participants at the time that they receive their outpatient appointment letter. This information will be provided in the form of the patient information sheet.Treatment decisions for SBD are made at the time of the ENT outpatient clinic. Therefore receiving this information before the outpatient appointment allows the parent/guardian adequate time to consider the study fully before they're asked whether or not they wish to participate. The participants being recruited are children too young to provide consent or assent; it is therefore important that the parents of the participants are well informed and have time to consider the information fully. Parents/guardians will be offered the opportunity to ask any questions that they may have at the time of the outpatient clinic and will also be made aware that participation is voluntary and can be withdrawn at any time. The consent form will be completed with the research psychologist to ensure that the parent/guardian is fully aware of what the trial involves and is therefore making an informed choice. The research psychologist has had training in mental capacity assessment and is competent in assessing and ensuring comprehension and reasoned decision making. If eligible the participant will be offered entry into the study and parents will provide informed consent at the time of their clinic attendance. This will avoid delay in the assessment or treatment process and is in line with the treatment format of the clinic.

Risks, burdens and benefits:

The investigators do not know what is the best course of treatment for young children with SDB. There is a single study of preschool age children with SDB with a low follow up rate (Biggs. PLoS One 2015). This study found no difference in cognitive development or behaviour at 3 years post diagnosis irrespective of whether the child had undergone adenotonsillectomy or not. These children had cognitive weakness compared to non-snoring controls, and this got worse whether they received surgical treatment or were just observed. Current practice of offering adenotonsillectomy may be subjecting children to a painful operation which offers them no long term benefit. Set against this, adenotonsillectomy is known to immediately improve quality of life in older children but it is not know if the difference seen at 7 months post randomisation is still present 2-3 years later if children have grown out of SDB. This study therefore has equipoise.

ELIGIBILITY:
Inclusion Criteria:

1. Aged more than 2 years 6 months and less than 5 years of age at time of recruitment
2. A diagnosis of SDB based on clinical criteria.
3. Enlarged tonsils on examination (2 or more on standard Brodsky scale)

Exclusion Criteria:

1. Recurrent tonsillitis as main symptoms leading to consideration for AT
2. Known genetic, cranio-facial or psychiatric condition likely to affect airway, cognition or behaviour
3. Obesity (Body Mass Index > 2.5 standard deviation from mean for age and gender)
4. Severe OSA (Apnoea Hypopnoea Index greater than 30 / hour on sleep study)
5. Severe chronic health conditions that may hamper participation. This may include severe congenital heart disease, cystic fibrosis, sickle cell anaemia, or poorly controlled epilepsy)
6. A history of significant hypertension (defined as greater than the 99th percentile (CDC prediction equations) plus 5mmHg for either systolic or diastolic.
7. Concurrent use of ADHD medicines, psychotropic medications (anti-depressants, anxiolytics, anti-psychotics), hypnotics or anti convulsants.
8. Previous adenotonsillectomy, tonsillectomy or adenoidectomy.
9. Receiving Continuous Positive Airway Pressure as a treatment
10. A parent or Guardian who is unable to read and thus understand the consent form.
11. A family planning to move out of the area within the next 9 months.
12. Severe snoring since birth.

Ages: 30 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2016-12; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Cognition | 8 months
  Weschler Pre-School and Primary Scale of Intelligence (WPPSI) The full Score IQ measures of each of the two groups will be compared at baseline (to ensure no group differences at the start) and again at the end of the study period. Any difference at the end of the study period will provide information to answer the key study question, and potentially to power a larger definitive study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Tremlett, BM, FRCA, Principal Investigator — South Tees Hospitals NHS FT
Locations (1):
- The James Cook University Hospital, Middlesbrough, Cleveland, United Kingdom

IPD SHARING:
Plan to Share IPD: No